CLINICAL TRIAL: NCT00656292
Title: Perioperative HMG-CoA-Reductase-Inhibitors: A Pilot Study Assessing the Role of "Statin" Therapy and Perioperative Inflammatory Response in Patients Undergoing Major Orthopedic Surgery
Brief Title: Assessing the Role of "Statin" Therapy and Perioperative Inflammatory Response in Patients Undergoing Major Orthopedic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael Brown, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-002881
Record Dates: First submitted 2008-04-04; First posted 2008-04-11 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Perioperative Inflammatory Response
Keywords: Plasma concentrations of inflammatory markers; C-Reactive Protein (CRP); Interleukin-6 (IL-6); Tumor Necrosis Factor-Alpha (TNF); Aspartate Aminotransferase (AST); Alanine Aminotransferase (ALT); Creatine Kinase (CK)
MeSH Terms: interventions — Simvastatin

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Simvastatin (Placebo Comparator): Subjects randomized to this arm will receive statin therapy (simvastatin 40 mg) two days before surgery -- allowing three doses of simvastatin before incision -- and these will be continued until patients are either discharged from the hospital or have completed a 3-day postoperative course (6 days of simvastatin therapy), whichever occurs earlier. If patients are unable to take oral medications, the enteral route via nasogastric tube (at our institution, nasogastric tubes are routinely placed for both lumbar and thoracic instrumentation) will be used to deliver either placebo or the statin, as no parenteral form of this drug is currently available.
  Interventions: Drug: Simvastatin
- Placebo (Experimental): Subjects randomized to this arm will receive placebo two days before surgery -- allowing three doses of placebo before incision -- and these will be continued until patients are either discharged from the hospital or have completed a 3-day postoperative course (6 days of placebo), whichever occurs earlier. If patients are unable to take oral medications, the enteral route via nasogastric tube (at our institution, nasogastric tubes are routinely placed for both lumbar and thoracic instrumentation) will be used to deliver either placebo or the statin, as no parenteral form of this drug is currently available.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — 40 mg po/nasogastric tube (NG) every day for 6 days
  Other Names: Zocor
  Arms: Simvastatin
Drug: Placebo — 1 pill po/NG every day x 6 days
  Arms: Placebo

SUMMARY:
The purpose of the present study is to quantify the degree of modulation, if any, in the perioperative inflammatory response associated with statins use. Specifically, we hypothesize that:

In a population of patients undergoing elective orthopedic spine surgery, administration of a specific statin (Simvastatin, Zocor®, Merck Pharmaceuticals), will be associated with a decrease in perioperative inflammatory markers when compared to patients not taking statins

DETAILED DESCRIPTION:
Previous studies have reported activation of the body's immune system during the perioperative period.1 Typically, this "stress response" is limited and goes unnoticed by the patient and health care team. However, physiologic insults that occur during major surgery may elicit a more pronounced response known as the systemic inflammatory response syndrome (SIRS). Such a response is of great clinical consequence, as it is known to significantly worsen perioperative morbidity and mortality.1 HMG Co-A Reductase Inhibitors (hereafter identified by the common name, "the statins") are potent inhibitors of cholesterol synthesis, and their role in the treatment of atherosclerosis and prevention of coronary artery disease is well documented.2-5 Interestingly, data from animal studies have shown that statins have unique anti-inflammatory properties that are independent of their lipid lowering effects.6 Recently, statin therapy has been associated with a reduced incidence of perioperative cardiovascular and neurologic complications in major vascular and thoracic surgery patients as well as improved outcomes in patients experiencing acute coronary syndrome (ACS).7-13 In all ACS patient populations studied, improvement in outcome has been attributed to coronary plaque stabilization, presumably a result of statins mitigating the local inflammatory response at the level of the coronary plaque.

The purpose of this study is to quantify the magnitude of perioperative inflammation during major orthopedic spine surgery and determine whether statins alter this systemic physiologic response.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for elective major spine surgery (multilevel (2-6 level) open thoracic or lumbar spine surgery with instrumentation)

Exclusion Criteria:

1. Pregnancy
2. Lactating females
3. Oral or parenteral corticosteroid use in the past 30 days
4. Elevation of AST or ALT > 3x normal
5. Elevation of creatinine kinase > 2x normal
6. Previous adverse drug reaction to any medication in the statin class
7. Current use of fibrates, niacin, itraconazole, ketoconazole, macrolide antibiotics, HIV protease inhibitors and/or nefazodone
8. Active liver disease
9. Current statin use
10. Anti-inflammatory use of the following medications within the last 30 days:

    * Sulfasalazine
    * Mycophenolate
    * Cyclosporine
    * Cyclophosphamide
    * Azathioprine
    * Chlorambucil
    * Minocycline
    * Myochrysine
    * Penicillamine
    * Hydroxychloroquine
    * Leflunomide
11. Any medications listed in 3 or 10 above in the post-operative period
12. Use of Activated protein C at any time during the patients hospitalization
13. Use of anti-inflammatory medications listed below within the last 30 days:

    * Leflunomide
    * Sulfasalazine
    * Mycophenolate
    * Cyclosporine
    * Cyclophosphamide
    * Azathioprine
    * Chlorambucil
    * Minocycline
    * Myochrysine
    * Penicillamine
    * Hydroxychloroquine
    * Methotrexate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Brown, M.D., Principal Investigator — Mayo Clinic Department of Anesthesiology; Daryl Kor, M.D., Principal Investigator — Mayo Clinic Department of Anesthesiolgy
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Simvastatin | Placebo
Started | 32 | 29
Completed | 29 | 24
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Screen failure | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin | Placebo | Total
Number analyzed (Participants) | 32 | 29 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (16.2) | 56.3 (15.6) | 55.6 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 16 | 38
  Male | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  United States | 32 | 29 | 61

OUTCOME MEASURES:

1. Primary Outcome: Median Concentration of Aspartate Aminotransferase (AST)
Description: Description: AST is an enzyme found in high amounts in liver, heart, and muscle cells. This test is mainly done along with other tests such as alkaline phosphatase and bilirubin to diagnose and monitor liver disease. This test evaluates hepatocyte integrity, as serum levels of this enzyme rise in response to a variety of forms of injury to hepatic cells. The normal range is 10 to 40 U/L.
Time Frame: baseline, at the start of the surgical procedure (0 hrs), 8 hrs, 24 hrs, 48 hrs, 72 hrs
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 29 | 24
U/L
  baseline | 24.5 [18.8 to 31.0] | 24.5 [21.0 to 27.8]
  time 0 hours | 21.0 [18.0 to 24.0] | 20.0 [17.0 to 24.0]
  time 8 hours | 29.0 [21.0 to 33.0] | 25.0 [19.3 to 31.5]
  time 24 hours | 41.5 [28.0 to 84.8] | 30.5 [22.5 to 72.5]
  time 48 hours | 53.0 [26.5 to 118.0] | 35.0 [25.8 to 80.8]
  time 72 hours | 56.5 [29.3 to 100.3] | 44.0 [28.0 to 97.5]

2. Secondary Outcome: Median Concentration of Alanine Aminotransferase (ALT)
Description: An enzyme normally present in liver and heart cells that is released into the bloodstream when the liver or heart is damaged. The blood ALT levels are elevated with liver damage (for example, from viral hepatitis) or with an insult to the heart (for example, from a heart attack). The normal range is 7 to 56 U/L.
Time Frame: baseline, at the start of the surgical procedure (0 hrs), 8 hrs, 24 hrs, 48 hrs, 72 hrs
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 29 | 24
U/L
  baseline | 23 [18.5 to 28.0] | 22.0 [17.5 to 28.5]
  time 0 hours | 16.5 [14.0 to 25.0] | 16.0 [14.0 to 24.0]
  time 8 hours | 18.0 [13.0 to 23.0] | 16.5 [12.3 to 21.0]
  time 24 hours | 20.5 [17.0 to 29.5] | 17.0 [12.7 to 23.5]
  time 48 hours | 23.0 [16.5 to 42.0] | 18.0 [14.80 to 25.0]
  time 72 hours | 24.0 [18.5 to 45.5] | 25.0 [16.0 to 39.0]

3. Secondary Outcome: Median Concentration of C-Reactive Protein (CRP)
Description: C-reactive protein (CRP) is a substance produced by the liver in response to inflammation. Normal CRP levels are below 3.0 mg/L.
Time Frame: baseline, at the start of the surgical procedure (0 hrs), 8 hrs, 24 hrs, 48 hrs, 72 hrs
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 29 | 24
mg/L
  baseline | 3.0 [3.0 to 3.5] | 3.0 [3.0 to 4.2]
  time 0 hours | 3.0 [3.0 to 3.2] | 3.0 [3.0 to 5.1]
  time 8 hours | 3.0 [3.0 to 5.2] | 4.1 [3.0 to 8.0]
  time 24 hours | 47.5 [22.8 to 70.6] | 52.5 [26.9 to 86.9]
  time 48 hours | 139.7 [112.7 to 199.2] | 157.8 [96.0 to 258.2]
  time 72 hours | 122.4 [100.3 to 173.1] | 197.2 [120.5 to 235.3]

4. Secondary Outcome: Median Concentration of Creatine Kinase (CK)
Description: A creatine kinase test may be used to detect inflammation of muscles or muscle damage due to muscle disorders. A person may have muscle injury with few or nonspecific symptoms, such as weakness, fever, and nausea, that may also be seen with a variety of other conditions. A healthcare practitioner may use a CK test to help detect muscle damage in these cases, especially if someone is taking a drug such as a statin. Normal values at rest are usually between 60 and 174 IU/L.
Time Frame: baseline, at the start of the surgical procedure (0 hrs), 8 hrs, 24 hrs, 48 hrs, 72 hrs
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 29 | 24
U/L
  baseline | 89.5 [58.5 to 112.5] | 111.0 [86.0 to 154.2]
  time 0 hours | 71.0 [51.0 to 134.8] | 103.0 [66.0 to 147.0]
  time 8 hours | 527.0 [213.0 to 754.0] | 257.0 [206.8 to 558.0]
  time 24 hours | 1345.0 [434.5 to 2621.2] | 647.0 [273.0 to 1688.0]
  time 48 hours | 973.0 [446.0 to 2724.0] | 685.0 [272.0 to 1357.0]
  time 72 hours | 597.0 [355.0 to 1839.0] | 886.0 [253.0 to 1565.0]

5. Secondary Outcome: Median Concentration of Interleukin-6 (IL-6)
Description: Interleukin-6 (IL-6) may be used to help evaluate a person who has a condition associated with inflammation, such as lupus or rheumatoid arthritis, or with infection, such as sepsis. It may also be used in the evaluation of diabetes or cardiovascular disease. IL-6 is a cytokine, a protein produced by immune cells that acts on other cells to help regulate and/or promote an immune response. It also stimulates the production of acute phase reactants, proteins that increase in the blood with conditions that cause inflammation or tissue injury. Circulating IL-6 can be found in the blood of normal individuals in the 1 pg/mL range, with slight elevations during the menstrual cycle, modest elevations in certain cancers (melanoma) (10 pg/mL), and large elevations after surgery (30-430 pg/mL).
Time Frame: baseline, at the start of the surgical procedure (0 hrs), 8 hrs, 24 hrs, 48 hrs, 72 hrs
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 29 | 24
ng/ml
  baseline | 1.5 [0.1 to 2.8] | 2.4 [0.7 to 3.8]
  time 0 hours | 1.2 [0.1 to 2.3] | 1.8 [0.5 to 3.4]
  time 8 hours | 50.0 [24.6 to 135.7] | 56.7 [27.8 to 135.7]
  time 24 hours | 64.2 [41.5 to 182.4] | 70.2 [51.9 to 172.7]
  time 48 hours | 89.2 [46.6 to 155.9] | 87.0 [39.3 to 175.7]
  time 72 hours | 37.7 [16.3 to 55.5] | 45.2 [22.0 to 92.4]

6. Secondary Outcome: Median Concentration of Tumor Necrosis Factor-Alpha (TNF)
Description: Tumor Necrosis Factor Alpha is a cell signaling protein (cytokine) involved in systemic inflammation and is one of the cytokines that make up the acute phase reaction. TNF is important to the body because it helps regulate the response of the immune system to a foreign object, especially to the present cancerous tumor. It promotes inflammation, produces other cells used in the inflammatory response, and can help cells heal. The normal range is 5 to 27.2 pg/ml.
Time Frame: baseline, at the start of the surgical procedure (0 hrs), 8 hrs, 24 hrs, 48 hrs, 72 hrs
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 29 | 24
pg/ml
  baseline | 1.0 [0.7 to 1.2] | 0.85 [0.6 to 1.3]
  time 0 hours | 0.95 [0.60 to 1.21] | 0.96 [0.71 to 1.30]
  time 8 hours | 0.94 [0.64 to 1.34] | 0.86 [0.54 to 1.06]
  time 24 hours | 1.25 [0.89 to 1.53] | 1.00 [0.67 to 1.26]
  time 48 hours | 1.57 [1.05 to 1.70] | 1.37 [0.89 to 1.63]
  time 72 hours | 1.58 [1.14 to 1.85] | 1.36 [0.99 to 1.69]

ADVERSE EVENTS:
Time Frame: 72 hours after spine surgery
Arm/Group | Simvastatin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/29 | 3/24
Other Adverse Events (participants affected / at risk) | 0/29 | 1/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=29) | Placebo (N=24)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Cardiac disorders) | 0 (0) | 1 (1)
Non-invasive ventilation required > 24 hrs post-op (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=29) | Placebo (N=24)
Post-op Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes